CLINICAL TRIAL: NCT04756583
Title: Advance Care Planning Notifications in General Inpatient Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00107026
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2023-01

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Notification system
- Control (No Intervention)

INTERVENTIONS:
Other: Notification system — Email and page notification sent to clinicians for patients at high-risk of mortality in 30 days and 6 months
  Arms: Intervention

SUMMARY:
This study will evaluate the impact of and response by physicians on Hospital Medicine/General Internal Medicine service to a notification identifying seriously ill patients at high risk of death within 30 days as well as within 6 months in a cluster randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Attending Physician on the Hospital Medicine or General Internal Medicine Service at Duke University Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of advance care planning notes as measured by electronic health record data during hospitalization | Up to 30 days

SECONDARY OUTCOMES:
Proportion of advance care planning codes billed as measured by electronic health record data | Up to 30 days
Proportion of Palliative Care Consults (Inpatient/Outpatient) as measured by electronic health record data | Up to 90 days
Proportion of patients discharged to hospice as measured by electronic health record data | Up to 30 days
Proportion of patients' code status changed to Do-Not-Resuscitate as measured by electronic health record data | Up to 30 days
Proportion of patient deaths as measured by electronic health record data | Up to 14 days
Proportion of patient deaths as measured by electronic health record data | Up to 30 days
Proportion of patient deaths as measured by electronic health record data | Up to 6 months
Proportion of patient re-admitted to the hospital as measured by electronic health record data | Up to 30 days
Proportion of patient re-admitted to the hospital as measured by electronic health record data | Up to 6 months
Proportion of advance care planning paperwork filed as measured by electronic health record data | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David Casarett, MD, Principal Investigator — Duke University; Jessica Ma, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No